CLINICAL TRIAL: NCT07301502
Title: A Randomized, Double-blind, Placebo-controlled, Dose-escalation Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Preliminary Efficacy of AK152 in Healthy Volunteers and Patients With Alzheimer' s Disease
Brief Title: A Clinical Trial of AK152 in Healthy Volunteers and Patients With Alzheimer' s Disease
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AK152-101
Record Dates: First submitted 2025-12-01; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer' s Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK152 regimen (Active Comparator)
  Interventions: Drug: AK152
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AK152 — Subjects receiving single or multiple doses of AK152 injection.
  Arms: AK152 regimen
Drug: Placebo — Subjects receiving single or multiple doses of placebo injection.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind phase I clinical trial to evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Preliminary Efficacy of AK152 in Healthy Volunteers and Patients with Alzheimer' s Disease.

DETAILED DESCRIPTION:
This is a randomized, double-blind phase I clinical trial to evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Preliminary Efficacy of AK152 in Healthy Volunteers and Patients with Alzheimer' s Disease. Subjects will be randomized to receive AK152 regimen or placebo treatment.

ELIGIBILITY:
Key Inclusion Criteria - Part 1 (Healthy Volunteers):

1. Healthy male or female subjects aged 18 to 40 years (inclusive) at the time of signing the informed consent form (ICF).
2. Body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females; body mass index (BMI) = weight (kg) / height² (m²) within the range of 19.0-26.0 kg/m² (inclusive).
3. Subjects agree to take protocol-specified contraception measures and refrain from donating sperm or oocytes from signing the ICF through the treatment period and for at least 90 days after the last administration of study drug; women of childbearing potential must be non-pregnant and non-lactating.
4. Subjects are able to understand and voluntarily sign a written ICF before any study-specific procedures are performed, and are able to comply with the study procedures and follow-up requirements.

Key Exclusion Criteria - Part 1 (Healthy Volunteers):

1. Known allergy to components of AK152 injection or any monoclonal antibody, or high risk of allergy.
2. History or presence of any systemic disease that may interfere with study results.
3. Clinically significant abnormalities in vital signs at screening or prior to randomization.
4. Clinically significant laboratory abnormalities at screening or prior to randomization per investigator judgment.
5. Use of any medication (including prescription, OTC, herbal medicines, dietary supplements) within 4 weeks before randomization or within 5 half-lives of the medication (whichever is longer), or planned use during the study.
6. History of frequent alcohol consumption within 24 weeks or inability to abstain during inpatient stay.
7. Drug abuse or positive urine drug screen at screening.
8. Smokers consuming >5 cigarettes/day within 12 weeks prior to screening or unable to abstain during the inpatient period.
9. Excessive intake of tea, coffee, or other caffeine-containing beverages.

Key Inclusion Criteria - Part 2 (Alzheimer' s Disease Patients):

1. Able to understand and voluntarily sign a written ICF before any study-specific procedures are performed, and able to comply with study procedures and follow-up requirements.
2. Aged 50 to 85 years (inclusive) at the time of signing the ICF.
3. BMI within 17.0-35.0 kg/m² (inclusive).
4. Subjects agree to take protocol-specified contraception measures and refrain from donating sperm or oocytes from signing the ICF through the treatment period and for at least 90 days after the last dose; women must be non-pregnant and non-lactating.
5. The subject must have an identified trial partner who must sign a separate ICF.
6. Meets the 2011 NIA-AA core clinical criteria for MCI due to AD or mild AD dementia.
7. Evidence of brain amyloid deposition confirmed by Aβ-PET/CT at screening.

Key Exclusion Criteria - Part 2 (Alzheimer' s Disease Patients):

1. History or evidence of malignancy involving any organ system within 5 years prior to screening, regardless of treatment or remission status (except completely cured carcinoma in situ of the cervix, non-metastatic squamous cell carcinoma of the skin, or basal cell carcinoma).
2. Severe or unstable disease at screening or prior to randomization that may affect study assessments.
3. Major neurological disorder (other than AD) that may affect cognition or ability to complete study procedures.
4. Transient ischemic attack (TIA) or stroke within 12 months prior to randomization.
5. Clinically significant abnormalities on brain MRI at screening.
6. Known allergy to components of AK152 injection or any monoclonal antibody, or high risk of allergy.
7. History of alcohol or drug abuse within 2 years prior to screening or prior to randomization.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) | Up to approximately 8 weeks after the last dose
  The incidence of AEs.

SECONDARY OUTCOMES:
Peak concentration (Cmax) | Up to approximately 8 weeks after the last dose
  Measure and assess the Cmax of AK152.
Time to peak (Tmax) | Up to approximately 8 weeks after the last dose
  Measure and assess the Tmax of AK152.
Area under the curve (AUC) | Up to approximately 8 weeks after the last dose
  Measure and assess the AUC of AK152.
Half-life (t1/2) | Up to approximately 8 weeks after the last dose
  Measure and assess the t1/2 of AK152.
Immunogenicity characteristics of AK152 | Up to approximately 8 weeks after the last dose
  Number and percentage of subjects with detectable anti-drug antibodies (ADA) and neutralizing antibodies (Nab) after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The Frist Affiliated Hospital of USTC, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No